CLINICAL TRIAL: NCT05694546
Title: Re-engagement at Discharge 2: Improving Post-hospital Outcomes for Adults With HIV in Zambia
Brief Title: Re-engagement at Discharge 2
Acronym: ReCharge2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University Teaching Hospital, Lusaka, Zambia (Other); University of Alabama at Birmingham (Other); University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Cassidy Claassen, Associate Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R34MH122265 (NIH)
Record Dates: First submitted 2022-01-07; First posted 2023-01-23 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: HIV/AIDS; Hospitalization; Transitions of Care; Opportunistic Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Opportunistic Infections

STUDY DESIGN:
Intervention Model Description: Community health worker follow-up after discharge from hospital
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community Health Worker Post-Discharge Intervention (Experimental): This group will be offered a community-based visit from a community health worker following hospital discharge.
  Interventions: Behavioral: Community Health Worker Post-Discharge Intervention

INTERVENTIONS:
Behavioral: Community Health Worker Post-Discharge Intervention — Clients will be offered a community-based follow-up from a community health worker after hospital discharge.

SUMMARY:
Early post-discharge mortality is high among Zambians living with HIV admitted to the hospital. This may be due to missed opportunities in post-discharge care, such as inadequate follow-up and treatment. In this study the investigators will develop and pilot a new approach to post-discharge HIV care to improve care coordination and treatment adherence.

DETAILED DESCRIPTION:
Many people living with HIV (PLHIV) have poor outcomes following hospitalization, including high mortality, readmission, and gaps in HIV care engagement. This is likely multi-factorial and not all etiologies may be modifiable. While high mortality may due to incurable cancer, the majority of deaths in PLHIV are thought to be caused by infectious diseases for which treatments exist. However, succumbing to these life-threatening infections after discharge may be due to poor understanding of discharge instructions, lack of post hospital care, and poor understanding of required follow up. Psychosocial support also plays a role in the mental and physical health of these sick patients.

In ReCharge 1, the investigators gathered formative data and identified at least three major factors that undermine HIV clinical outcomes after hospital discharge. First, there are gaps in continuity of care between the discharging facility and outpatient. Second, support from family is often suboptimal due to lack of understanding on the cause of illness, lack of HIV status disclosure, and the cost of care. Third, HIV comorbidities may underpin or complicate the immediate reason for discharge or the post-discharge engagement in care. These data were disseminated to local experts in Zambia including from the Ministry of Health and used to create a new care model for post-discharge HIV care. The care model draws from other successful programs in Zambia. In ReCharge 2 the investigators now propose to pilot the program and assess feasibility, acceptability, and potential for clinical impact.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years
* HIV-positive
* Hospitalized for at least 1 night at study site
* Clinically stable and expected to be discharged according to their clinician
* Objective evidence of suboptimal HIV outcome, defined as HIV viral load above the lower limit of the assay or T-cell cluster of differentiation 4 count <=200.

Exclusion Criteria:

* Unable to provide informed consent
* No phone
* Planning to reside outside of Lusaka urban district after discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cassidy Claassen, MD, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- Zambia (2):
  - Levy Mwanawasa University Teaching Hospital, Lusaka
  - University Teaching Hospital, Lusaka

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Community Health Worker Post-Discharge Intervention
Started | 97
Completed | 86
Not Completed | 11
Not completed — Lost to Follow-up | 11

BASELINE CHARACTERISTICS:
Arm/Group | Community Health Worker Post-Discharge Intervention
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 97
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Zambia | 97
CD4 <200 [Count of Participants; unit: Participants] | 84

OUTCOME MEASURES:

1. Primary Outcome: Post-Discharge Visits
Description: Proportion of discharged patients who are successfully visited after discharge.
Time Frame: Through three months post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Community Health Worker Post-Discharge Intervention
Number analyzed (Participants) | 97
Participants | 92

2. Primary Outcome: Comprehensive Post-Discharge Visits
Description: Number of participants that receive a comprehensive discharge follow-up visit from a community health worker
Time Frame: Through three months post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Community Health Worker Post-Discharge Intervention
Number analyzed (Participants) | 97
Participants | 67

3. Primary Outcome: Post-Discharge Clinic Visits
Description: Proportion of initial post-discharge visits to the HIV clinic that are attended by the participant's community health worker
Time Frame: Through three months post-discharge
Reporting Status: Not Posted

4. Secondary Outcome: HIV Viral Load Suppression
Description: Proportion of clients with suppressed HIV viral load at 6 months post-discharge.
Time Frame: 6 months post-discharge
Reporting Status: Not Posted

5. Secondary Outcome: Mortality
Description: Proportion of clients alive at 6 months post-discharge.
Time Frame: 6 months post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Community Health Worker Post-Discharge Intervention
Number analyzed (Participants) | 97
Participants
  Confirmed Alive | 77
  Confirmed Dead | 19
  Lost to Follow Up | 1

6. Secondary Outcome: Retention in HIV Care
Description: Retention in HIV care after discharge defined by no gap of >28 days off antiretroviral therapy from discharge date to 6 months post-discharge date
Time Frame: 6 months post-discharge
Reporting Status: Not Posted

7. Secondary Outcome: Antiretroviral Therapy Clinic Visit
Description: Antiretroviral therapy clinic visit within 1 month of discharge
Time Frame: 1 month post-discharge
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: No difference
Arm/Group | Community Health Worker Post-Discharge Intervention
All-Cause Mortality (participants affected / at risk) | 19/97
Serious Adverse Events (participants affected / at risk) | 28/97
Other Adverse Events (participants affected / at risk) | 0/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Community Health Worker Post-Discharge Intervention (N=97)
Hospital Readmission (Surgical and medical procedures) | 28 — Readmission to hospital

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT05694546/Prot_SAP_ICF_000.pdf